CLINICAL TRIAL: NCT06165913
Title: The Evaluation of Facial Bone Changes After Early Implant Placement Protocols "Clinically and Radiographically".
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Ahmed Ali Abdelkader Radwan, principle investigator, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1993
Record Dates: First submitted 2023-11-29; First posted 2023-12-12 (Actual); Last update posted 2023-12-12 (Actual); Status verified 2023-12

CONDITIONS: Bone Loss; Dental Implants
Keywords: facial bone loss; early implant placement; bone changes after implant
MeSH Terms: conditions — Bone Diseases, Metabolic

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group (1): Early implant placement(type II) group. (Experimental): Patients will be scheduled for tooth extraction then performing implant placement between 4-8 weeks later after soft tissue healing.
  Interventions: Procedure: Early implant placement(type II)
- Group (2): Early implant placement (type III) group. (Experimental): Patients will be scheduled for tooth extraction and performing implant placement between 12-16 weeks with partial bone healing.
  Interventions: Procedure: Early implant placement (type III)

INTERVENTIONS:
Procedure: Early implant placement(type II) — in group 1, Tooth extraction will be performed with care to preserve alveolar bone walls. After 4-8 weeks from tooth extraction, dental implant will be placed
  Arms: Group (1): Early implant placement(type II) group.
Procedure: Early implant placement (type III) — in group 2, Tooth extraction will be performed with care to preserve alveolar bone walls. After 12-16 weeks from tooth extraction, dental implant will be placed.
  Arms: Group (2): Early implant placement (type III) group.

SUMMARY:
The loss of a single tooth could negatively impact the physiologic occlusion because of the tipping of neighboring teeth and the super-eruption of the opposing teeth. In addition, it compromises the esthetic, especially when anterior teeth are missing, leading to psychological problems such as loss of confidence and avoidance of smiling in public with a defect in phonetics.

Restoration of the missing tooth is achieved in many ways, including removable dental appliances, fixed dental prostheses and dental implants.

Implant placement is classified into different protocols according to the time of placement in relation to the time of extraction. These different protocols are immediate implant placement (type 1) on the day of extraction; early implant placement (type 2) after 4-8 weeks with soft tissue healing; early implant placement (type 3) after 12-16 weeks with partial bone healing; and delayed dental implant placement (type 4) after complete bone healing at least 6 months after tooth extraction the Aim of the work: to evaluate facial bone changes after early implant placement protocols clinically and radiographically.

DETAILED DESCRIPTION:
Dental implant is the most reliable option as it replace the natural tooth without affecting the neighboring teeth and preserve the surrounding tooth structure with better functional performance. Implant placement is classified in different protocols according to the time of placement in relation to time of extraction. These Different protocols are immediate implant placement (type 1) on the day of extraction, early implant placement (type 2) after 4-8 weeks with soft tissue healing, early implant placement (type 3) after 12-16 weeks with partial bone healing and delayed dental implant placement (type 4) after complete bone healing at least after 6 months from tooth extraction.

Early Implant placement (type 2) after 4-8 weeks post extraction that allows soft tissue healing, resolution of local pathology, shorter treatment time, increase soft tissue volume makes it easier to manipulate the surgical flaps and enables flap advancement for primary closure.

Early implant placement (type 3) after 12-16 weeks with partial bone healing allow more implant stability than in type 1 and type 2 implant placement. The soft tissues are usually completely recovered, enabling tension free closure of the flap and improves esthetic outcomes. However, bone remodeling is more advanced. Perimplant defects may still be present, but with partial bone healing they are reduced in dimension.

Aim of the Work:

The evaluation of facial bone changes after early implant placement protocols clinically and radiographically.

ELIGIBILITY:
Inclusion Criteria:

1. Patients above 20 years old.
2. Patients with hopeless tooth in the maxillary anterior premolar region with socket type I indicated for extraction due to failure endodontic treatment, vertical root fracture, …etc.
3. Patients in good health with no medical contra-indication that would prevent routine oral surgery.
4. Patients with a positive attitude towards oral hygiene

Exclusion Criteria:

1. Patients with relevant medical conditions that may delay healing or compromise implant osseointegration.
2. Presence of risk factors as diabetes or smoking.
3. Pregnant or lactating women.
4. Absence of buccal bone after tooth extraction.
5. Insufficient vertical inter-arch space to accommodate the prostheses.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2023-05-30 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
The pocket depth will be measured by mm | 6-12 months
  the effect of type of implant placement in G1and G2 will be evaluated clinically regarding pocket depth. pocket depth will be measured by mm these measurements will be done after 6 and 12 months post dental implant placement.
primary radiographical outcome | 12 months
  the effect of type of implant placement in G1and G2 will be evaluated radiographically by cone beam computed tomography (CBCT) regarding facial bone loss.
  CBCT will be taken 24 hours after surgery (base line) and 12 months from surgery to obtain following measurement:
  A. Vertical facial bone length (VFBL) is the perpendicular distance from implant platform (0) to most coronal point of the facial bone.
primary radiographical outcome | 12 months
  the effect of type of implant placement in G1and G2 will be evaluated radiographically by cone beam computed tomography (CBCT) regarding facial bone loss.
  CBCT will be taken 24 hours after surgery (base line) and 12 months from surgery to obtain following measurement:
  B. Horizontal facial bone thickness (HFBT) is the thickness of facial bone in anterior-posterior direction in respect to implant fixture: Horizontal bone thickness will be measured at margin of platform level 0,1,2and3 mm from implant platform level.

SECONDARY OUTCOMES:
The Plaque index | 6-12 months
  The effect of type of implant placement in G1and G2 will be evaluated clinically regarding Plaque index
The Bleeding on probing | 6-12 months
  The effect of type of implant placement in G1and G2 will be evaluated clinically regarding Bleeding on probing.
Horizontal bone thickness will be measured at the middle and apex of implant fixture | 12 months
  the effect of type of implant placement in G1and G2 will be evaluated radiographically by cone beam computed tomography (CBCT) regarding facial bone loss.
  CBCT will be taken 24 hours after surgery (base line) and 12 months from surgery to obtain following measurement:
  • Horizontal bone thickness will be measured at the middle and apex of implant fixture.

CONTACTS AND LOCATIONS:
Overall Officials: Rehab F Ghouraba, PHD, Study Director — Tanta University
Locations (1):
- Tanta University faculty of dentistry, Tanta, Egypt

IPD SHARING:
Plan to Share IPD: No